CLINICAL TRIAL: NCT03740659
Title: Aqueous Humour Concentrations After Topical apPlication of combinEd Levofloxacin-dexamethasone Eye dRops and of Its Single Components: a randoMized, assEssor-blinded, Parallel-group Study in Patients Undergoing Cataract Surgery - iPERME
Brief Title: Evaluation Of Aqueous Humor Of Levofloxacin-Dexamethasone Eye Drops And Of Its Components In Patients Undergoing Cataract Surgery
Acronym: iPERME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NTC srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LevoDesa_05-2017
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Levofloxacin; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A randomized, assessor-blinded, parallel-group study.
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Levofloxacin + Dexamethasone (Experimental): Levofloxacin 5 mg/ml + Dexamethasone 1 mg/ml (30 μl administered twice before Limbal paracentesis).
  Limbal paracentesis will be performed prior to cataract surgery.
  Interventions: Drug: Levofloxacin + Dexamethasone
- Levofloxacin (Active Comparator): Levofloxacin 5 mg/ml (30 μl administered twice before Limbal paracentesis).
  Limbal paracentesis will be performed prior to cataract surgery.
  Interventions: Drug: Levofloxacin
- Dexamethasone (Active Comparator): Dexamethasone 1.14 mg/ml (26 μl administered twice before Limbal paracentesis).
  Limbal paracentesis will be performed prior to cataract surgery.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Levofloxacin + Dexamethasone — Levofloxacin + Dexamethasone ophthalmic solution + dexamethasone 21-phosphate administered twice: 90(±15) min. and 60(±15) min. before limbal paracentesis.
  Arms: Levofloxacin + Dexamethasone
Drug: Levofloxacin — Levofloxacin ophthalmic solution (Oftaquix®) administered twice: 90 (±15) min. and 60 (±15) min. before limbal paracentesis).
  Other Names: Oftaquix®
  Arms: Levofloxacin
Drug: Dexamethasone — Dexamethasone ophthalmic solution (Tamesad®) administered twice: 90 (±15) min. and 60 (±15) min. before Limbal paracentesis.
  Other Names: Tamesad®
  Arms: Dexamethasone

SUMMARY:
The purpose of this study is to evaluate the penetration of levofloxacin and dexamethasone 21-phosphate into the aqueous humour after ocular administration in combination or as single active ingredients.

DETAILED DESCRIPTION:
In most cases, postoperative care after cataract surgery consists of antiinflammatory and antibacterial drug therapy. The use of an ophthalmic solution containing the combination of a steroid and an antibiotic is routinely used in clinical practice; however, treatment duration could favour the emergence of antibiotic resistance. The study treatment associating a broad-spectrum antibiotic with a highly effective corticosteroid that can be used for a short period of time (one week) is therefore of considerable interest.

The aim of this study is to measure the concentrations of levofloxacin and dexamethasone in the aqueous humour after topical application of the combined ophthalmic solution and its single components.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female patients, aged ≥40 years
3. Patient undergoing phacoemulsification
4. Corneal thickness between 450 μm and 600 μm as measured by means of pachymetry
5. Corneal integrity confirmed by means of fluorescein test
6. Adequate pupil dilation assessed at screening
7. Female patients of childbearing potential must have a negative pregnancy test
8. Ability to fully understand all study procedures

Exclusion Criteria:

1. Corneal epithelium integrity not confirmed by fluorescein test
2. History of corneal disease or dystrophy
3. History of ocular trauma with corneal damage
4. History of acute ocular inflammation (including uveitis) in the 6 months prior to screening
5. Previous ocular surgery (including laser treatment)
6. Glaucoma
7. Treatment with an ophthalmic investigational drug in the 3 months prior to screening
8. Treatment with any topical ocular drug within 12 hours before start of cataract surgery other than study drugs and instillation of topical anaesthetic within 10 minutes before start of surgery
9. Treatment with any topical steroid or antibiotic drug in the 7 days prior to cataract surgery
10. Treatment with any systemic steroid or antibiotic drug in the 7 days prior to cataract surgery
11. Known hypersensitivity to levofloxacin, other fluoroquinolones or dexamethasone
12. Pregnant or lactating women
13. Patients who have received any investigational drug during the preceding 30 days or 5 times the plasma half-life, or who have previously participated in this trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Nardi, Prof., Principal Investigator — A.O.U. Pisana - P.O. di Cisanello
Locations (2):
- Italy (2):
  - ASST Santi Paolo e Carlo di Milano - P.O. San Paolo di Milano, Milan, MI
  - A.O.U. Pisana - P.O. di Cisanello, Pisa, PI

REFERENCES:
- [Derived] Figus M, Posarelli C, Romano D, Nardi M, Rossetti L. Aqueous humour concentrations after topical apPlication of combinEd levofloxacin-dexamethasone eye dRops and of its single components: a randoMised, assEssor-blinded, parallel-group study in patients undergoing cataract surgery: the iPERME study. Eur J Clin Pharmacol. 2020 Jul;76(7):929-937. doi: 10.1007/s00228-020-02863-7. Epub 2020 Apr 13. PMID 32285142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period:
  * Date of first enrolment: 4 September 2018
  * Date study finalized (last patient last visit): 6 December 2018
  Study centres:
  * U.O. Oculistica Universitaria, Azienda Ospedaliera Universitaria Pisana, Presidio Ospedaliero di Cisanello, Pisa;
  * Clinica Oculistica, Presidio Ospedale San Paolo, Milan.
Pre-assignment Details: Planned sample size n.120; randomized patients n.125; screened patients n.133 (1 patient screened for both eyes).
Groups:
- Levofloxacin + Dexamethasone: Levofloxacin 0.5% + DSP 0.132% (w/v) eye drops (TEST product). One ml contains levofloxacin hemihydrate 5.12 mg, corresponding to 5 mg of levofloxacin, and DSP 1.32 mg, corresponding to 1 mg of dexamethasone.
  Administration route: ocular instillation
  Dose and regimen: two 30 μl doses 30 minutes apart, one 90 ± 15 minutes prior to surgery and the other 60 ± 15 minutes prior to surgery (each dose contains 150 μg anhydrous levofloxacin and 39.6 μg DSP).
- Levofloxacin: Levofloxacin 0.5% eye drops (Oftaquix®). One ml contains 5,12 mg of levofloxacin hemihydrate equal to 5 mg of levofloxacin.
  Administration route: ocular instillation
  Dose and regimen: two 30 μl doses 30 minutes apart, one 90 ± 15 minutes prior to surgery and the other 60 ± 15 minutes prior to surgery (each dose contains 150 μg anhydrous levofloxacin).
- Dexamethasone: Dexamethasone sodium phosphate 0.15% eye drops (Tamesad®). One ml contains 1.5 mg of DSP corresponding to 1.14 mg/ml of dexamethasone.
  Administration route: ocular instillation
  Dose and regimen: two 26 μl doses 30 minutes apart, one 90 ± 15 minutes prior to surgery and the other 60 ± 15 minutes prior to surgery (each dose containing 39 μg DSP).
Period: Overall Study
Arm/Group | Levofloxacin + Dexamethasone | Levofloxacin | Dexamethasone
Started | 42 | 42 | 41
Completed | 42 | 42 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Main eligibility criteria included patients of both genders, aged ≥40 years and scheduled for phacoemulsification.
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin + Dexamethasone | Levofloxacin | Dexamethasone | Total
Number analyzed (Participants) | 42 | 42 | 41 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 6 | 17
  >=65 years | 35 | 38 | 35 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.45 (7.60) | 75.38 (8.38) | 74.59 (8.00) | 74.14 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 21 | 69
  Male | 15 | 21 | 20 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 42 | 40 | 40 | 122
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 42 | 42 | 41 | 125

OUTCOME MEASURES:

1. Primary Outcome: Aqueous Humour Concentration of Levofloxacin
Description: Defined as the concentration of levofloxacin into the aqueous humour in all the three arms: Levofloxacin + Dexamethasone, Dexamethasone and Levofloxacin.The concentration of levofloxacin has been measured by LC tandem mass spectrometry.
Time Frame: 90±15 min after the first administration of the study treatments
Population: Participants in all Arms/Groups were assessed for this Outcome Measure regardless of treatment type
Measure: Mean (95% Confidence Interval); unit: nmol/mL
Arm/Group | Levofloxacin + Dexamethasone | Levofloxacin | Dexamethasone
Number analyzed (Participants) | 42 | 42 | 41
nmol/mL | 1.970 [1.648 to 2.292] | 2.151 [1.708 to 2.594] | 0 [0 to 0]

2. Primary Outcome: Aqueous Humour Concentration of Dexamethasone 21-phosphate
Description: Defined as the concentration of dexamethasone 21-phosphate into the aqueous humour in all the three arms: Levofloxacin + Dexamethasone, Dexamethasone and Levofloxacin. The concentration of dexamethasone 21-phosphate has been measured by LC tandem mass spectrometry.
Time Frame: 90±15 min after the first administration of the study treatments
Population: Participants in all Arms/Groups were assessed for this Outcome Measure regardless of treatment type
Measure: Mean (95% Confidence Interval); unit: nmol/mL
Arm/Group | Levofloxacin + Dexamethasone | Levofloxacin | Dexamethasone
Number analyzed (Participants) | 42 | 42 | 41
nmol/mL | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Primary Outcome: Aqueous Humour Concentration of Dexamethasone
Description: Defined as the concentration of dexamethasone into the aqueous humour in all the three arms: Levofloxacin + Dexamethasone, Dexamethasone and Levofloxacin.The concentration of dexamethasone has been measured by LC tandem mass spectrometry.
Time Frame: 90±15 min after the first administration of the study treatments
Population: Participants in all Arms/Groups were assessed for this Outcome Measure regardless of treatment type
Measure: Mean (95% Confidence Interval); unit: nmol/mL
Arm/Group | Levofloxacin + Dexamethasone | Levofloxacin | Dexamethasone
Number analyzed (Participants) | 42 | 42 | 41
nmol/mL | 0.030 [0.025 to 0.035] | 0 [0 to 0] | 0.042 [0.035 to 0.048]

ADVERSE EVENTS:
Time Frame: From baseline to the study completion, approximately 2 hours
Arm/Group | Levofloxacin + Dexamethasone | Levofloxacin | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levofloxacin + Dexamethasone (N=42) | Levofloxacin (N=42) | Dexamethasone (N=41)
Mild Mydriasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03740659/Prot_SAP_000.pdf